CLINICAL TRIAL: NCT02062177
Title: Propofol Administered by Gastroenterologists by Target Controlled Infusion Pump During Endoscopy: a Randomized Double Blind Controlled Study
Brief Title: Propofol Administered by Gastroenterologists by Target Controlled Infusion Pump During Endoscopy
Acronym: Propofol TCI
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Università Vita-Salute San Raffaele (Other)
Responsible Party: Principal Investigator, Testoni Pier Alberto, Professor, Università Vita-Salute San Raffaele
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Propofol TCI endoscopy
Record Dates: First submitted 2014-02-03; First posted 2014-02-13 (Estimated); Results first posted 2014-09-08 (Estimated); Last update posted 2014-09-08 (Estimated); Status verified 2014-08

CONDITIONS: Sedation; Endoscopy
MeSH Terms: interventions — Propofol; Midazolam

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- propofol group (Experimental): 70 patients (35 upper endoscopy - 35 colonoscopy)
  Interventions: Drug: Propofol
- midazolam group (Active Comparator): 70 patients (35 upper endoscopy - 35 colonoscopy)
  Interventions: Drug: Midazolam

INTERVENTIONS:
Drug: Propofol — 70 patients (35 upper endoscopy - 35 colonoscopy) are sedated with propofol TCI (Target Controlled Infusion) pump (concentration 1.2-1.6 mcg/ml).
  Arms: propofol group
Drug: Midazolam — 70 patients (35 upper endoscopy - 35 colonoscopy) in group midazolam are sedated with midazolam 0.04 mg/Kg if aged < 70, 0.03 mg/Kg if aged > 70.
  Arms: midazolam group

SUMMARY:
Many studies address safety of non-anesthesiologist propofol sedation (NAPS) for gastrointestinal endoscopy. Target Controlled Infusion (TCI) is a sophisticated tool for providing optimal sedation regimen and avoiding under or oversedation. The objective of the study is to compare standard moderate sedation during upper endoscopy and colonoscopy versus propofol NAPS.

ELIGIBILITY:
Inclusion Criteria:

* age < 18 years
* American Society of Anesthesiologists risk I-II
* patients undergoing to Gastroscopy or Colonoscopy

Exclusion Criteria:

* significant systemic disease
* allergic reactions to any of study drugs
* chronic use of opioids or psychiatric disorders
* pregnancy
* Mallampati score > 2
* age < 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2014-02; Primary Completion 2014-02 (Actual); Study Completion 2014-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pier Alberto Testoni, Professor, Study Director — Vita-Salute San Raffalele University- San Raffaele Hospital
Locations (1):
- San Raffaele Hospital, Milan, Italy, Italy

REFERENCES:
- [Derived] Fanti L, Gemma M, Agostoni M, Rossi G, Ruggeri L, Azzolini ML, Dabizzi E, Beretta L, Testoni PA. Target Controlled Infusion for non-anaesthesiologist propofol sedation during gastrointestinal endoscopy: The first double blind randomized controlled trial. Dig Liver Dis. 2015 Jul;47(7):566-71. doi: 10.1016/j.dld.2015.03.003. Epub 2015 Mar 14. PMID 25840875

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 140 consecutive outpatients were scheduled to undergo Upper Endoscopy (70 patients) or complete Colonoscopy (70 patients) from 17 th February 2014 to 5 th May 2014 in Endoscopy Unit of San Raffaele Hospital - Milan.
Pre-assignment Details: Exclusion criteria were: significant systemic disease (ASA III-IV), allergic reactions to study drugs, chronic use of opioids, psychiatric disorders, pregnancy, difficult airways (Mallampati score >2), age <18 years.
  A gastroenterology attending fellow (GF), not directly involved in the procedure, provided sedation.
Groups:
- Propofol Group: A total amount of 70 patients (35 undergoing upper endoscopy + 35 undergoing colonoscopy) were sedated with propofol TCI (Target Controlled Infusion) pump. Target concentration was initially set at 1.2-1.6 µg/ml according to patient's body weight and general condition.
  35 patients of the group undergoing colonoscopy received also iv fentanyl (1μg/Kg) for pain control.
- Midazolam Group: A total amount of 70 patients (35 undergoing upper endoscopy + 35 undergoing colonoscopy) were sedated with midazolam (0.04 mg/kg if aged <70 years - 0.03 mg/kg if aged >70 years).
  35 patients of the group undergoing colonoscopy received also iv fentanyl (1μg/Kg) for pain control.
Period: Overall Study
Arm/Group | Propofol Group | Midazolam Group
Started | 70 | 70
Completed | 70 | 70
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Propofol Group: 70 patients (35 undergoing upper endoscopy + 35 undergoing colonoscopy) were sedated with propofol TCI (Target Controlled Infusion) pump. Target concentration was initially set at 1.2-1.6 µg/ml according to patient's body weight and general condition.
  35 patients of the group undergoing colonoscopy received also iv fentanyl (1μg/Kg) for pain control.
  Patients in this group received placebo boluses with normal saline to warrant blindness to the randomization group of both patient and endoscopist. (because of the well-known difference in the physical appearance of the study drugs, to maintain blindness of endoscopist, a fabric curtain was drawn across patient's arm covering the i.v. line and TCI pump).
- Midazolam Group: 70 patients (35 undergoing upper endoscopy + 35 undergoing colonoscopy) were sedated with midazolam (0.04 mg/kg if aged <70 years - 0.03 mg/kg if aged >70 years).
  35 patients of the group undergoing colonoscopy received also iv fentanyl (1μg/Kg) for pain control.
- Total: Total of all reporting groups
Arm/Group | Propofol Group | Midazolam Group | Total
Number analyzed (Participants) | 70 | 70 | 140
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 55 | 57 | 112
  >=65 years | 15 | 13 | 28
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 32 | 62
  Male | 40 | 38 | 78
Region of Enrollment [Number; unit: participants]
  Italy | 70 | 70 | 140

OUTCOME MEASURES:

1. Primary Outcome: Endoscopist's Satisfaction (Visual Analog Scale) About Sedation
Description: Visual Analog Scale from 0 to100 (0=dissatisfaction - 100=complete satisfaction) will be used to assess the technical difficulty of examination and the satisfaction with sedation of patient experienced by endoscopist
Time Frame: at the end of the exam
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Propofol Group; n=35, 35 | Midazolam Group; n=35, 35
Number analyzed (Participants) | 70 | 70
units on a scale
  upper endoscopy | 93 (14) | 83 (21)
  colonoscopy | 98 (11) | 87 (12)

2. Primary Outcome: Patient's Satisfaction (Visual Analog Scale) About Sedation Before Discharge
Description: When completely awake, patients will be asked to rate the degree of pain/discomfort and the degree of satisfaction about quality of sedation from 0 to100 (0=dissatisfaction - 100=complete satisfaction)
Time Frame: before discharge
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Propofol Group; n=35, 35 | Midazolam Group; n=35, 35
Number analyzed (Participants) | 70 | 70
units on a scale
  Upper endoscopy | 94 (18) | 76 (25)
  Colonoscopy | 95 (9) | 85 (14)

3. Primary Outcome: Patient's Satisfaction (Visual Analog Scale) About Sedation 24-72 Hours After Procedure
Description: Patients will be contacted by telephone 24-72 hours after discharge and asked about their satisfaction about the quality of sedation, rated on a verbal rating scale, from 0 to 100 (0=dissatisfaction; 100=complete satisfaction)
Time Frame: at 24-72 hours after procedure
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Propofol Group; n=35, 35 | Midazolam Group; n=35, 35
Number analyzed (Participants) | 70 | 70
units on a scale
  Upper endoscopy | 93 (20) | 77 (27)
  Colonoscopy | 97 (9) | 88 (16)

4. Secondary Outcome: Time (Minutes) to Dischargeability of Patient From Endoscopic Unit
Description: After endoscopy, patients will be transferred to recovery area and evaluated every 5 minutes until they will be ready to be discharged from the Endoscopy Unit. Recovery will be assessed using the Modified Aldrete Scoring System; patients will be considered fit for discharge with a Modified Aldrete Scoring System score of 18 or more, stable vital signs and without nausea, vomiting, or itching.
Time Frame: one day
Reporting Status: Not Posted

5. Secondary Outcome: Number of Participants With Adverse Events as a Measure of Safety
Description: Number of patients with adverse events (hypotension, bradycardia, hypoxemia,...)
Time Frame: one day
Reporting Status: Not Posted

ADVERSE EVENTS:
Description: Serious and other (non serious) adverse events were not collected
Groups:
- Propofol Group; n=35, 35; Midazolam Group; n=35, 35: 35 upper endoscopy 35 colonoscopy
Arm/Group | Propofol Group; n=35, 35 | Midazolam Group; n=35, 35
Serious Adverse Events (participants affected / at risk) | 0/70 | 0/70
Other Adverse Events (participants affected / at risk) | 0/70 | 0/70

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No